CLINICAL TRIAL: NCT02730429
Title: ENGOT-EN3-NSGO/PALEO: A Randomized, Double-blind, Placebo-controlled, Phase II Trial of Palbociclib in Combination With Letrozole Versus Placebo in Combination With Letrozole for Patients With Estrogen Receptor Positive Advanced or Recurrent Endometrial Cancer.
Brief Title: Trial of Letrozole + Palbociclib/Placebo in Metastatic Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Gynecologic Cancer Intergroup (GCIG) (Other); North Eastern German Society of Gynaecological Oncology (Other); Multicenter Italian Trials in Ovarian cancer and gynecologic malignancies (MITO) (Unknown); Grupo Español de Investigación en Cáncer de Ovario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENGOT-EN3-NSGO/PALEO
Record Dates: First submitted 2016-01-14; First posted 2016-04-06 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letrozole + placebo (Placebo Comparator): letrozole 2.5mg once daily days 1-28 every 28 days shall be administered until progression of disease or unacceptable toxicity. Letrozole is administered as standard of care in both study arms.
  Placebo for palbociclib once daily days 1-21 every 28 days shall be administered until progression of disease or unacceptable toxicity.
  Interventions: Drug: Letrozole
- Letrozole + palbociclib (Experimental): Palbociclib 125mg once daily days 1-21 every 28 days shall be administered until progression of disease or unacceptable toxicity.
  letrozole 2.5mg once daily days 1-28 every 28 days shall be administered until progression of disease or unacceptable toxicity.
  Letrozole is administered as standard of care in both study arms.
  Interventions: Drug: Palbociclib/placebo; Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib/placebo — Palbociclib or a placebo is administered together with standard of care letrozole
  Arms: Letrozole + palbociclib
Drug: Letrozole — Letrozole is standard of care in both arms

SUMMARY:
This randomized double-blind, placebo-controlled phase 2 trial is evaluating superiority of Letrozole-palbociclib combination versus letrozole-placebo combination in ER positive endometrioid adenocarcinoma of endometrium

DETAILED DESCRIPTION:
This multicenter, prospective, randomized, double-blind, placebo-controlled phase 2 study is evaluating the efficacy of letrozole-palbociclib combination against letrozole-placebo combination in women with ER+ advanced or relapsed endometrial cancer.

Stratification

Patients are stratified according to:

1. Number of prior lines of therapy (primary advanced disease vs. 1st relapse vs. ≥2 relapses)
2. Measurable vs. evaluable disease
3. Prior use of MPA/Megace

Randomization 1:1 randomization The patients with prior MPA/Megace treatment will be capped to a maximum of 50%.

Study arms

Patients are randomized to one of the two treatment arms:

* Arm A: (comparator) letrozole-placebo combination therapy until progression.
* Arm B: (experimental arm): Letrozole- palbociclib combination therapy until progression

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmed endometrial cancer of endometrioid type. Mixed tumor histology is allowed if the non-endometrioid component is less than 5%. Tumor must be estrogen receptor positive.
2. Patients may have received adjuvant chemotherapy for stage 1 or 2.
3. Patients may have received any lines of chemotherapy for primary advanced (stage 3-4) or relapsed disease.
4. Patients may have received external beam radiotherapy, brachytherapy, and surgery.
5. Patient may have received maximum one line of endocrine therapy containing MPA/Megace only.
6. Patients must have measureable disease or evaluable disease on CT scan according to RECIST 1.1 outside irradiated field.
7. Patients must give informed consent
8. Patients must have a WHO performance status of 0-1
9. Patients must have an adequate bone-marrow, renal and hepatic function
10. Life expectancy of at least 12 weeks
11. Patients must be fit to receive combination therapy
12. Patient's age >18 years
13. Patient is post-menopausal. Patients under the age of 55 with intact ovaries shall undergo hormonal verification.
14. Patients with preserved reproductive capacity must have a negative pregnancy test (β-HCG test in urine or serum) prior to commencing study treatment

Exclusion Criteria:

1. Non-endometrioid adenocarcinomas, sarcomas, small cell carcinoma with neuroendocrine differentiation or non-epithelial cancers.
2. Previous anti-cancer endocrine therapy other than MPA/Megace. This means that eg. tamoxifen is not allowed prior to study entry.
3. Concurrent cancer therapy
4. Previous treatment with Palbociclib or other CDK inhibitors.
5. Concurrent treatment with an investigational anticancer agent or participation in another anticancer clinical trial within 21 days before entering into study.
6. Treatment within 21 days prior to randomization with any investigational drug, radiotherapy,
7. Major injuries or surgery within the past 21 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
8. Previous malignant disease, except patients with other malignant disease, for which the patient has been disease-free for at least three years. Concurrent other malignant disease except for curatively treated carcinoma in situ of the cervix or basal cell carcinoma of the skin.
9. Active infection or other serious underlying medical condition, which might prevent the patient from receiving treatment or to be followed.
10. Evidence of significant medical illness, abnormal laboratory finding or psychiatric illness/social situation that would, in the Investigator's judgment, makes the patient inappropriate for this study.
11. Known uncontrolled hypersensitivity to the investigational drugs.
12. History of major thromboembolic event defined as:
13. History of a cerebral vascular accident, transient ischemic attack or subarachnoid hemorrhage within the past 3 months.
14. History of clinically significant hemorrhage in the past 3 months.
15. Uncontrolled and/or symptomatic CNS metastasis or leptomeningeal carcinomatosis (dexamethasone/prednisone therapy will be allowed if administered as stable dose for at least one month prior randomization).
16. Significant cardiovascular diseases, including uncontrolled hypertension, uncontrolled clinically relevant cardiac arrhythmia, unstable angina or myocardial infarction within 6 months prior to randomization, congestive heart failure > NYHA III, severe peripheral vascular disease, clinically significant pericardial effusion.
17. Pregnancy or breastfeeding. Patients with preserved reproductive capacity, unwilling to use a medically acceptable method of contraception for the duration of the trial and for 3 months afterwards.
18. Active or chronic hepatitis C and/or B infection
19. Persistence of clinically relevant grade 3-4 therapy related toxicity from previous chemo and/or radiotherapy
20. Known hypersensitivity to the trial drugs, or to their excipients.
21. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
22. Unable or unwilling to swallow tablets/capsules

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS). Increase in median PFS in experimental arm versus comparator arm | 26 months
  To be measured (in months) and reported

SECONDARY OUTCOMES:
PFS of patients in the sub-populations as described under stratification factors. Increase in median PFS in experimental arm versus comparator arm | 26 months
  To be measured (in months) and reported
Overall Response Rate (ORR) according to RECIST | 26 months
  To be measured (in %) and reported
Disease Control Rate (DCR) for at least 12 weeks | 26 months
  To be measured (in %) and reported
Time to First Subsequent Therapy (TFST) | 36 months
  TFST: time from randomization to first subsequent therapy or death. To be measured (in months) and reported
Progression-Free Survival 2 (PFS2) | 48 months
  PFS2: time from randomization to second objective disease progression or death. To be measured (in months) and reported
Time to Second Subsequent Therapy (TSST) | 48 months
  TSST: time from randomization to second subsequent therapy or death.To be measured (in months) and reported
Patient Reported Outcomes (PROs) like Quality of Life questionnaire EORTC-QLQ-C30 & EORTC-QLQ-EN24 | 48 months
  These are the validated questionnaires to be answered by patients. Results to be reported as descriptive and on a scale of 1-10
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 48 months
  To be reported on %
Compliance in the two treatment arms. | 48 months
  Missed dosages in both arm will be reported.
Dose reductions/interruptions in the two treatment arms | 48 months
  To be reported on %

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor R Mirza, MD, Study Chair — NSGO
Locations (1):
- NSGO-CTU, Copenhagen, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
As all endpoints are matured, the individual participant data will be shared.

REFERENCES:
- [Derived] Mirza MR, Bjorge L, Marme F, Christensen RD, Gil-Martin M, Auranen A, Ataseven B, Rubio MJ, Salutari V, Luczak AA, Runnebaum IB, Redondo A, Lindemann K, Trillsch F, Ginesta MPB, Roed H, Kurtz JE, Petersson KS, Nyvang GB, Sehouli J. Palbociclib plus letrozole in estrogen receptor-positive advanced/recurrent endometrial cancer: Double-blind placebo-controlled randomized phase II ENGOT-EN3/PALEO trial. Gynecol Oncol. 2025 Jan;192:128-136. doi: 10.1016/j.ygyno.2024.12.003. Epub 2024 Dec 9. PMID 39657575